CLINICAL TRIAL: NCT01610531
Title: COPARIME: Pilot Study of a Target Detection of Malignant Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BRD/10/11-N
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-05

CONDITIONS: Patients at Risk for Melanoma
Keywords: Cohort; Melanoma; targeted screening; risks function; cost effectiveness
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: SAMScore questionnaire — Patients assessed at high risk according to the SAMScore

SUMMARY:
Melanoma is nowadays an important public health problem because its growing incidence. Mass screening for melanoma is not recommended worldwide because of its low cost-effectiveness. Nevertheless targeted screening for patients at high risk for melanoma is promoted. This study is designed to assess the effectiveness and the acceptability of a melanoma targeted screening of melanoma, to estimate the risk function to develop a melanoma among patients at high risk according to the SAMScore and to estimate the ratio cost/ efficacy of the melanoma targeted screening. A cohort of 7700 patients is carried out in 2 departments covered by a registry of cancers. The recruitment had began in April 2011. Patients assessed at high risk according to the SAMScore were proposed a skin examination by their GP every year.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years old,
* consulting their GP,
* assessed at risk for melanoma according to the SAMScore
* signed the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4118 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Prevalence ratios between those of the COPARIME cohort and those of the general population. | 5 years
  Number of melanomas detected / Number of patients at high risk of melanoma defined by our selection tool.

SECONDARY OUTCOMES:
Probability to develop a melanoma at one year. | 1 years
Cost ratio for a screened melanoma. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel NGUYEN, Doctor, Study Chair — Nantes University Hospital
Locations (1):
- University Hospital, Nantes, France

REFERENCES:
- [Derived] Rat C, Hild S, Gaultier A, Khammari A, Bonnaud-Antignac A, Quereux G, Dreno B, Nguyen JM. Anxiety, locus of control and sociodemographic factors associated with adherence to an annual clinical skin monitoring: a cross-sectional survey among 1000 high-risk French patients involved in a pilot-targeted screening programme for melanoma. BMJ Open. 2017 Oct 5;7(10):e016071. doi: 10.1136/bmjopen-2017-016071. PMID 28982813
- [Derived] Rat C, Grimault C, Quereux G, Dagorne M, Gaultier A, Khammari A, Dreno B, Nguyen JM. Proposal for an annual skin examination by a general practitioner for patients at high risk for melanoma: a French cohort study. BMJ Open. 2015 Jul 29;5(7):e007471. doi: 10.1136/bmjopen-2014-007471. PMID 26224016
- [Derived] Rat C, Quereux G, Grimault C, Gaultier A, Khammari A, Dreno B, Nguyen JM. Melanoma incidence and patient compliance in a targeted melanoma screening intervention. One-year follow-up in a large French cohort of high-risk patients. Eur J Gen Pract. 2015 Jun;21(2):124-30. doi: 10.3109/13814788.2014.949669. Epub 2014 Aug 20. PMID 25141184